CLINICAL TRIAL: NCT02391688
Title: Evaluation of the Potential Pharmacokinetic Interactions Between Probe Drugs in the Geneva Phenotyping Cocktail
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jules Desmeules (Other)
Responsible Party: Sponsor-Investigator, Jules Desmeules, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-061
Record Dates: First submitted 2015-02-19; First posted 2015-03-18 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Drug Interaction
MeSH Terms: interventions — Caffeine; Omeprazole; Flurbiprofen; Dextromethorphan; Midazolam; Bupropion; fexofenadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Experimental): Oral intake of:
  caffeine 50 mg dextromethorphan 10 mg omeprazole 10 mg flurbiprofen 10 mg midazolam 1 mg
  Interventions: Drug: Caffeine, omeprazole, flurbiprofen, dextromethorphan, midazolam
- Treatment B (Experimental): Oral intake of:
  fexofenadine 25 mg
  Interventions: Drug: Fexofenadine
- Treatment C (Experimental): Oral intake of:
  bupropion 20 mg
  Interventions: Drug: Bupropion
- Treatment D (Experimental): Oral Intake of Geneva cocktail (A+B+C):
  caffeine 50 mg dextromethorphan 10 mg omeprazole 10 mg flurbiprofen 10 mg midazolam 1 mg fexofenadine 25 mg bupropion 20 mg
  Interventions: Drug: Caffeine, omeprazole, flurbiprofen, dextromethorphan, midazolam; Drug: Bupropion; Drug: Fexofenadine

INTERVENTIONS:
Drug: Caffeine, omeprazole, flurbiprofen, dextromethorphan, midazolam
  Arms: Treatment A; Treatment D
Drug: Bupropion
  Arms: Treatment C; Treatment D
Drug: Fexofenadine
  Arms: Treatment B; Treatment D

SUMMARY:
Phenotyping is an approach largely used for the evaluation of the activity of cytochromes and transporters in vivo. It consists of the administration of probe substances metabolised by a specific cytochrome or transported by P-glycoprotein (P-gp) for example, followed by the determination of a metabolic ratio or the evaluation of the plasmatic or urinary concentrations of the probe substances. The administration of a cocktail containing several probe substances allows the simultaneous evaluation of the activity of several cytochromes and P-gp in a single test.

When a cocktail approach is used it is important to make sure that no drug-drug interactions occur between the probes within the cocktail. The validation of the lack of interactions, which is the aim of the study, consists of demonstrating that there is no difference in the pharmacokinetic parameters and/or metabolic ratios when a probe is administered alone or as part of the cocktail. The Geneva cocktail consists of caffeine, bupropion, flurbiprofen, omeprazole, dextromethorphan, midazolam and fexofenadine for the simultaneous phenotyping of CYP1A2, CYP2B6, CYP2C9, CAP2C19, CYP2D6, CYP3A4 and P-gp, respectively.

Probe and metabolite concentrations will be measured in capillary blood using a dried blood spot (DBS) analysis. To further facilitate sampling, a new simple device will be used to ensure the precision of capillary blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged from 18 to 60 years
* BMI between 18 and 27
* Understanding of French language and able to give a written inform consent.

Exclusion Criteria:

* smoker
* pregnant women
* taking drugs which alter cytochrome P450 (CYP) activity
* renal or hepatic impairment
* medical history of chronic alcoholism or abuse of psychoactive drugs
* liver transplantation
* sensitivity to any of the drugs used
* Alteration of hepatic tests, more than 2x normal (aspartate transaminase >100U/L ; alanine transaminase >100 units/L ; gamma-glutamyl transferase >80 units/L ; bilirubin >50µmol/L)
* Presenting genetic polymorphism of poor CYP2C9, CYP2C19, CYP2D6 metabolizer

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Area under the capillary blood concentration-time curve (AUC) of caffeine | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post treatment A or D
  Comparison of caffeine AUC when treatment A or D is administered
Area under the capillary blood concentration-time curve (AUC) of dextromethorphan | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post treatment A or D
  Comparison of dextromethorphan AUC when treatment A or D is administered
Area under the capillary blood concentration-time curve (AUC) of flurbiprofen | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post treatment A or D
  Comparison of flurbiprofen AUC when treatment A or D is administered
Area under the capillary blood concentration-time curve (AUC) of midazolam | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post treatment A or D
  Comparison of midazolam AUC when treatment A or D is administered
Area under the capillary blood concentration-time curve (AUC) of omeprazole | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post treatment A or D
  Comparison of omeprazole AUC when treatment A or D is administered
Area under the capillary blood concentration-time curve (AUC) of fexofenadine | 0, 0.5, 1, 2, 3, 4, 6, 8 hours post treatment B or D
  Comparison of fexofenadine AUC when treatment B or D is administered
Area under the capillary blood concentration-time curve (AUC) of bupropion | 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post treatment C or D
  Comparison of bupropion AUC when treatment C or D is administered

SECONDARY OUTCOMES:
Metabolic ratio (MR) of paraxanthine blood concentration /caffeine blood concentration | 0.5, 1, 2, 3, 4, 6, 8 hours post treatment A or D
  Comparison of paraxanthine/caffeine MRs between treatment A and D
Metabolic ratio (MR) of dextrorphan blood concentration /dextromethorphan blood concentration | 0.5, 1, 2, 3, 4, 6, 8 hours post treatment A or D
  Comparison of dextrorphan/dextromethorphan MRs between treatment A and D
Metabolic ratio (MR) of 4-hydroxyflurbiprofen blood concentration /flurbiprofen blood concentration | 0.5, 1, 2, 3, 4, 6, 8 hours post treatment A or D
  Comparison of 4-hydroxyflurbiprofen/flurbiprofen MRs between treatment A and D
Metabolic ratio (MR) of 1-hydroxymidazolam blood concentration /midazolam blood concentration | 0.5, 1, 2, 3, 4, 6, 8 hours post treatment A or D
  Comparison of 1-hydroxymidazolam/midazolam MRs between treatment A and D
Metabolic ratio (MR) of 5-hydroxyomeprazole blood concentration /omeprazole blood concentration | 0.5, 1, 2, 3, 4, 6, 8 hours post treatment A or D
  Comparison of 5-hydroxyomeprazole/omeprazole MRs between treatment A and D
Metabolic ratio (MR) of 4-hydroxybupropion blood concentration /bupropion blood concentration | 0.5, 1, 2, 3, 4, 6, 8, 12, 24 hours post treatment C or D
  Comparison of 4-hydroxybupropion/bupropion MRs between treatment C and D
Number of adverse events | at each drug administration day

OTHER OUTCOMES:
Correlation of drug concentrations (ng/ml) in DBS obtained with two sampling techniques for all administered drugs | 0.5, 1, 2, 3, 4, 6, 8 hours post treatment A, B, C and D

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Recherche Clinique, HUG, Rue Gabrielle Perret-Gentil 4, Geneva, Switzerland